CLINICAL TRIAL: NCT02194062
Title: A Comparison of Budesonide Nasal Irrigation in Different Head Positions and Fluticasone Nasal Spray in Post-operative Functional Endoscopic Sinus Surgery Patients With Chronic Rhinosinusitis With Nasal Polyposis
Brief Title: Comparison of Nasal Steroids After FESS in CRSwNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1407014259
Record Dates: First submitted 2014-07-15; First posted 2014-07-18 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-01

CONDITIONS: Sinusitis; Nasal Polyps
Keywords: Chronic rhinosinusitis with polyps; Nasal steroids; Functional endoscopic sinus surgery; SNOT-22; Lund-Kennedy
MeSH Terms: conditions — Sinusitis; Nasal Polyps | interventions — Fluticasone; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- fluticasone nasal spray (Active Comparator): Group one will be prescribed fluticasone nasal spray ( to use 2-50 mcg sprays to each nostril two times per day)
  Interventions: Drug: fluticasone nasal spray
- budesonide respule in head upright (Active Comparator): Group two will be prescribed budesonide respules (0.5 mg/2mL) to instill into each nostril in the upright position two times per day
  Interventions: Drug: Budesonide head upright
- budesonide head forward (Active Comparator): Group three will be prescribed budesonide respules (0.5 mg/2mL) to use instill into each nostril in the head forward position two times per day with their head angled downwards by having their head lean forward off the side of a bed.
  Interventions: Drug: Budesonide head forward

INTERVENTIONS:
Drug: fluticasone nasal spray — use 2-50 mcg sprays to each nostril two times per day
  Other Names: fluticasone propionate nasal; Flonase
  Arms: fluticasone nasal spray
Drug: Budesonide head upright — (0.5 mg/2mL) to instill into each nostril in the upright position two times per day
  Other Names: budesonide; pulmicort respules
  Arms: budesonide respule in head upright
Drug: Budesonide head forward — (0.5 mg/2mL) to instill into each nostril in the head forward position two times per day
  Other Names: budesonide; pulmicort respules
  Arms: budesonide head forward

SUMMARY:
The purpose of this study is to compare intranasal fluticasone spray with budesonide nasal saline rinses in both the upright and head forward positions in patients who have had functional endoscopic sinus surgery (FESS) for chronic rhinosinusitis with nasal polyposis (CRSwNP) and measure differences in Sinonasal Outcome Test-22 (SNOT-22) scores and Lund- Kennedy scores on rigid nasal endoscopy at time points 1 week, 3 weeks, 6 weeks, 2 months, 4 months, and 6 months post-op.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is an inflammatory condition of the lining of the nose and sinuses that lasts 12 weeks or longer with objective evidence of mucosal inflammation (1). CRSwNP is characterized by the presence of bilateral nasal polyps in the middle meatus. Patients with CRSwNP for whom medical therapy has failed, often have functional endoscopic sinus surgery.

Nasal steroids are important post-operatively to prevent polyps from recurring. Many studies have shown that nasal steroids are superior to placebo in maintaining improvement in symptom scores, such as SNOT-22, post-operatively by preventing polyps from returning (2). Nasal steroids can reduce inflammation locally and can prevent disease relapse without the systemic effects of oral steroids. However, there is no consensus as to which nasal steroid and which delivery method is most effective in treating these patients. Traditional nasal sprays, such as fluticasone spray, may not deliver the medication widely in the nasal cavity. Budesonide is available in a respule form that can be used to instill the medication in the nose. In an attempt to more effectively deliver the medication, changes in patient's head position has been prescribed to achieve better delivery (3). The safety of intranasal budesonide, a more potent steroid than fluticasone, has been established (4, 5). However, any improved efficacy over fluticasone nasal spray remains anecdotal as head to head comparisons have not previously been performed.

Practice patterns among rhinologists in the post-operative prescription of nasal steroids vary widely. Determining which medication/delivery method is more effective will help rhinologists better treat their patients and prevent symptoms, for which the surgery was performed, from returning.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have had FESS for CRSwNP within the study period

Exclusion Criteria:

1. Patients who are under the age of 18
2. Concurrent oral corticosteroid use of the equivalent of greater than 10 mg of prednisone use per day
3. The use of medications that accelerate the clearance of systemic cortisol (Dilantin, rifampin, amphetamines, and lithium)
4. The use of medications that inhibit the clearance of systemic cortisol (ketoconazole, amphotericin B, bupropion, fluoroquinolones)
5. Known hypersensitivity to corticosteroids
6. A personal history of Wegener's Granulomatosis or other autoimmune disease with nasal manifestations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Peter Manes, MD, Principal Investigator — Yale University School of Medicine, Asst Professor
Locations (2):
- United States (2):
  - Yale Physicians Bldg, New Haven, Connecticut
  - Yale ENT Stratford, Stratford, Connecticut

REFERENCES:
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Background] Snidvongs K, Kalish L, Sacks R, Sivasubramaniam R, Cope D, Harvey RJ. Sinus surgery and delivery method influence the effectiveness of topical corticosteroids for chronic rhinosinusitis: systematic review and meta-analysis. Am J Rhinol Allergy. 2013 May-Jun;27(3):221-33. doi: 10.2500/ajra.2013.27.3880. PMID 23710959
- [Background] Beule A, Athanasiadis T, Athanasiadis E, Field J, Wormald PJ. Efficacy of different techniques of sinonasal irrigation after modified Lothrop procedure. Am J Rhinol Allergy. 2009 Jan-Feb;23(1):85-90. doi: 10.2500/ajra.2009.23.3265. PMID 19379619
- [Background] Bhalla RK, Payton K, Wright ED. Safety of budesonide in saline sinonasal irrigations in the management of chronic rhinosinusitis with polyposis: lack of significant adrenal suppression. J Otolaryngol Head Neck Surg. 2008 Dec;37(6):821-5. PMID 19128710
- [Background] Sachanandani NS, Piccirillo JF, Kramper MA, Thawley SE, Vlahiotis A. The effect of nasally administered budesonide respules on adrenal cortex function in patients with chronic rhinosinusitis. Arch Otolaryngol Head Neck Surg. 2009 Mar;135(3):303-7. doi: 10.1001/archoto.2008.555. PMID 19289711
- [Derived] Neubauer PD, Schwam ZG, Manes RP. Comparison of intranasal fluticasone spray, budesonide atomizer, and budesonide respules in patients with chronic rhinosinusitis with polyposis after endoscopic sinus surgery. Int Forum Allergy Rhinol. 2016 Mar;6(3):233-7. doi: 10.1002/alr.21688. Epub 2015 Dec 17. PMID 26679480

RESULTS

PARTICIPANT FLOW:
Groups:
- Budesonide Respule in Head Upright: Group two will be prescribed budesonide respules (0.5 mg/2mL) to instill into each nostril in the upright position two times per day
  Budesonide: (0.5 mg/2mL) to instill into each nostril in the upright position two times per day
- Budesonide Head Forward: Group three will be prescribed budesonide respules (0.5 mg/2mL) to use instill into each nostril in the head forward position two times per day with their head angled downwards by having their head lean forward off the side of a bed.
  Budesonide: (0.5 mg/2mL) to instill into each nostril in the head forward position two times per day
Period: Overall Study
Arm/Group | Fluticasone Nasal Spray | Budesonide Respule in Head Upright | Budesonide Head Forward
Started | 10 | 10 | 12
Completed | 8 | 8 | 7
Not Completed | 2 | 2 | 5
Not completed — Lost to Follow-up | 2 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Nasal Spray | Budesonide Respule in Head Upright | Budesonide Head Forward | Total
Number analyzed (Participants) | 10 | 10 | 12 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 12 | 32
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (1) | 44.8 (1) | 39.6 (1) | 43.9 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 5 | 4 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 12 | 32
asthma [Number; unit: participants]
  yes | 5 | 5 | 5 | 15
  no | 5 | 5 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: SNOT-22 Scores
Description: SNOT22 is a validated scale which measures sinonasal symptoms for sinusitis patients. The 22 questions are rated on a scale of 0-5 for a maximum total score of 110. Higher scores represent more symptomatic patients.
Time Frame: 6 months post-op.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fluticasone Nasal Spray | Budesonide Respule in Head Upright | Budesonide Head Forward
Number analyzed (Participants) | 8 | 8 | 7
units on a scale | 31.5 [28.35 to 34.65] | 10.29 [9.59 to 10.99] | 15.88 [13.78 to 17.98]

2. Secondary Outcome: Lund-Kennedy Scoring for Nasal Endoscopy
Description: The Lund Kennedy scoring system for nasal endoscopy rates the severity of the sinusitis based on the endoscopic appearance of the nasal mucosa. Edema, secretions and the presence of polyps are rated from 0-2, for a total maximum score of 6 per each side of the nose. Higher scores represent more severe disease.
Time Frame: 6 months post-op
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fluticasone Nasal Spray | Budesonide Respule in Head Upright | Budesonide Head Forward
Number analyzed (Participants) | 8 | 8 | 7
units on a scale | 2.69 [2.06 to 3.30] | 0.5 [0.25 to 0.74] | 1.13 [0.71 to 1.54]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 6 months
Description: No difference in definitions for adverse events.
Groups:
- Fluticasone Group: Fluticasone nasal spray ( to use 2-50 mcg sprays to each nostril two times per day)
- Budesonide Respule in Head Upright: Budesonide respules (0.5 mg/2mL) to instill into each nostril in the upright position two times per day
- Budesonide Head Forward: budesonide respules (0.5 mg/2mL) to use instill into each nostril in the head forward position two times per day with their head angled downwards by having their head lean forward off the side of a bed.
Arm/Group | Fluticasone Group | Budesonide Respule in Head Upright | Budesonide Head Forward
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/12

LIMITATIONS AND CAVEATS:
Small numbers recruited due to time constraints. Not all patients included in final data analysis because of loss to follow up and time constraints of collecting the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No